CLINICAL TRIAL: NCT01859949
Title: Long Term Study Of Pnu-180307 For Short Children Born Small For Gestational Age (Sga) Without Epiphyseal Closure (Extension Of The Study 307-met-0021-002)
Brief Title: Long Term Study of Genotropin (Somatropin) for Short Children Born Small for Gestational Age (SGA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENASG-0021-007; A6281225 (Other: Alias Study Number); 2015-004552-21 (EudraCT Number)
Record Dates: First submitted 2013-04-17; First posted 2013-05-22 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-03

CONDITIONS: Short Stature Born Small for Gestational Age (SGA)
Keywords: Genotropin(somatropin); SGA; Short Stature; Long-term; Safety
MeSH Terms: conditions — Dwarfism | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genotropin (somatropin) (Experimental)
  Interventions: Drug: Genotropin (somatropin)

INTERVENTIONS:
Drug: Genotropin (somatropin) — Genotropin(somatoropin) 12 mg, Genotropin(somatropin) will be given at a dose of 0.067 mg/kg/day or 0.033 mg/kg/day to all participating patients

SUMMARY:
To assess the long-term safety of Genotropin(somatropin) on Small for Gestational Age (SGA) without epiphyseal closing.

ELIGIBILITY:
Inclusion Criteria:

Children with short stature due to SGA who received treatment in the study GENASG-0021-002.

Exclusion Criteria:

* Children who have any chronic disease requiring treatment with steroid hormone that may affect growth promotion including estrogen, androgen, anabolic hormone, and corticosteroids (except those for external use), and have received the treatment.
* Children who have received radiotherapy or chemotherapy.
* Children who have serious cardiac disease, renal disease, or hepatic disease.
* Children who have diabetes mellitus with a manifestation of abnormal glucose metabolism.
* Children who have serious chronic disease.
* Children who have malignant tumor.
* Children who are allergic to m-cresol.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2002-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- Japan (19):
  - University of Occupational and Environmental Health Hospital, Kitakyushu, Fukuoka
  - Gunma University Hospital, Maebashi, Gunma
  - Hiroshima City Hospital, Hiroshima, Hiroshima
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Hokkaido Social Service Association Obihiro Hospital, Obihiro, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Iwate Medical University Hospital, Morioka, Iwate
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka Medical Center and Research Institute for Maternal and Child Health, Izumi, Osaka
  - Osaka Employees' Pension Hospital, Osaka, Osaka
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Federal Officers' Mutual Aid Association Toranomon Hospital, Minato-ku, Tokyo
  - National Center for Child Health and Development, Setagaya-ku, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - Yamanashi University Hospital, Chūō, Yamanashi

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=GENASG-0021-007&StudyName=Long%20Term%20Study%20of%20Genotropin%20%28Somatropin%29%20for%20Short%20Children%20Born%20Small%20for%20Gestational%20Age%20%28SGA%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Before enrolled this study, participants with short stature due to SGA had completed the 1-year(12-month) treatment in previous study.
  Out of 62 participants who were enrolled this study, 61 participants were treated.
Groups:
- Dose-Increasing Group: Participants who were treated with somatropin 0.033 mg/kg/day in previous study for 12 months received a dose of 0.067 mg/kg/day
- Dose-Remaining Group: Participants who were treated with somatropin 0.067 mg/kg/day in previous study for 12 months were maintained on the same dose
Period: Overall Study
Arm/Group | Dose-Increasing Group | Dose-Remaining Group
Started | 29 (Treated participants) | 32 (Treated participants)
Completed | 15 | 15
Not Completed | 14 | 17
Not completed — Family Matters | 0 | 1
Not completed — Physician Decision | 2 | 4
Not completed — Withdrawal by Subject | 11 | 10
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-Increasing Group | Dose-Remaining Group | Total
Number analyzed (Participants) | 29 | 32 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.20 (1.64) | 5.40 (1.27) | 5.31 (1.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Month 12 (at the end of previous study) to 156
Population: Full Analysis Set (FAS) included participants who received at least 1 dose of study medication and had at least one observation after enrollment of this study.
Measure: Number; unit: participant
Arm/Group | Dose-Increasing Group | Dose-Remaining Group
Number analyzed (Participants) | 29 | 32
participant
  AE | 27 | 31
  SAE | 10 | 5

2. Secondary Outcome: Height Velocity Standard Deviation Score (SDS) for Chronological Age
Description: Height velocity is the yearly height gain. Height velocity SDS is calculated as following formula; Height velocity SDS = (height velocity - mean) / standard deviation,
  where mean and standard deviation were based on standard Japanese values of the participants age and gender.
  The scores were centred around zero. Negative score indicated a participant was smaller for their age/gender.
Time Frame: Month 12 (at the end of previous study) to 156
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Dose-Increasing Group | Dose-Remaining Group
Number analyzed (Participants) | 29 | 32
SDS
  Month 12 to 24 (Increasing: n=28, Remaining: n=32) | 2.782 (1.978) | 2.595 (1.731)
  Month 24 to36 (Increasing:n=26, Remaining:n=28) | 1.812 (1.526) | 1.696 (2.111)
  Month 36 to 48 (Increasing: n=24, Remaining: n=23) | 1.480 (1.543) | 0.824 (1.527)
  Month 48 to 60 (Increasing: n=21, Remaining: n=20) | -0.041 (2.081) | 0.480 (1.651)
  Month 60 to 72 (Increasing: n=20, Remaining: n=16) | -0.293 (1.585) | -0.046 (2.434)
  Month 72 to 84 (Increasing: n=15, Remaining: n=16) | -0.488 (3.117) | -1.511 (2.692)
  Month 84 to 96 (Increasing: n=11, Remaining: n=14) | 0.263 (1.802) | -0.114 (1.964)
  Month 96 to 108 (Increasing: n=9, Remaining: n=8) | 0.521 (2.058) | -0.466 (2.055)
  Month 108 to 120 (Increasing: n=6, Remaining: n=6) | -0.668 (2.126) | -0.590 (2.693)
  Month 120 to 132 (Increasing: n=5, Remaining: n=4) | -1.080 (1.953) | 1.173 (3.042)
  Month 132 to 144 (Increasing: n=4, Remaining: n=2) | 2.655 (4.329) | 0.730 (2.022)
  Month 144 to 156 (Increasing: n=3, Remaining: n=0) | 3.373 (1.995) | NA (NA) — Zero participants analyzed at this time point.

3. Secondary Outcome: Height Velocity
Description: Height velocity is the yearly height gain
Time Frame: Month 12 (at the end of previous study) to 156
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Dose-Increasing Group | Dose-Remaining Group
Number analyzed (Participants) | 29 | 32
cm/year
  Month 12 to 24 (Increasing: n=28, Remaining: n=32) | 7.83 (1.33) | 7.70 (1.19)
  Month 24 to 36 (Increasing: n=26, Remaining: n=28) | 6.88 (0.94) | 6.75 (1.52)
  Month 36 to 48 (Increasing: n=24, Remaining: n=23) | 6.68 (0.98) | 6.08 (1.14)
  Month 48 to 60 (Increasing: n=21, Remaining: n=20) | 6.06 (1.49) | 6.30 (1.24)
  Month 60 to 72 (Increasing: n=20, Remaining: n=16) | 6.08 (1.45) | 6.49 (1.37)
  Month 72 to 84 (Increasing: n=15, Remaining: n=16) | 4.89 (2.18) | 4.88 (1.86)
  Month 84 to 96 (Increasing: n=11, Remaining: n=14) | 5.16 (1.20) | 4.82 (2.12)
  Month 96 to 108 (Increasing: n=9, Remaining: n=8) | 5.18 (2.16) | 5.55 (2.42)
  Month 108 to 120 (Increasing: n=6, Remaining: n=6) | 5.72 (2.24) | 5.03 (1.86)
  Month 120 to 132 (Increasing: n=5, Remaining: n=4) | 4.84 (1.30) | 4.30 (1.84)
  Month 132 to 144 (Increasing: n=4, Remaining: n=2) | 4.38 (1.10) | 2.60 (0.14)
  Month 144 to 156(Increasing: n=3, Remaining: n=0) | 3.10 (1.92) | NA (NA) — Zero participants analyzed at this time point.

4. Secondary Outcome: Height SDS for Chronological Age
Description: Height SDS is calculated as following formula; Height SDS = (height - mean) / standard deviation,
  where mean and standard deviation were based on standard Japanese values on the participant age and gender.
  The scores were centred around zero. Negative score indicated a participant was smaller for their age/gender.
Time Frame: Month 12 (at the end of previous study) to 156
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Dose-Increasing Group | Dose-Remaining Group
Number analyzed (Participants) | 29 | 32
SDS
  Month 12 (Increasing: n=29, Remaining: n=32) | -2.53 (0.92) | -2.17 (0.96)
  Month 24 (Increasing: n=28, Remaining: n=32) | -2.02 (0.97) | -1.70 (1.03)
  Month 36 (Increasing: n=26, Remaining: n=28) | -1.80 (0.99) | -1.53 (1.10)
  Month 48 (Increasing: n=24, Remaining: n=23) | -1.48 (1.05) | -1.49 (1.15)
  Month 60 (Increasing: n=21, Remaining: n=20) | -1.53 (1.06) | -1.44 (1.10)
  Month 72 (Increasing: n=20, Remaining: n=16) | -1.56 (1.11) | -1.43 (1.06)
  Month 84 (Increasing: n=15, Remaining: n=16) | -1.73 (1.13) | -1.58 (1.17)
  Month 96 (Increasing: n=11, Remaining: n=14) | -1.52 (0.89) | -1.87 (1.36)
  Month 108 (Increasing: n=9, Remaining: n=8) | -1.52 (1.01) | -1.63 (1.48)
  Month 120 (Increasing: n=6, Remaining: n=6) | -1.52 (1.20) | -1.25 (0.59)
  Month 132 (Increasing: n=5, Remaining: n=4) | -1.96 (1.11) | -0.98 (0.51)
  Month 144 (Increasing: n=4, Remaining: n=2) | -1.73 (0.87) | -0.70 (0.42)
  Month 156 (Increasing: n=3, Remaining: n=0) | -1.77 (0.76) | NA (NA) — Zero participants analyzed at this time point.

5. Secondary Outcome: Height Velocity SDS for Bone Age
Description: To measure bone age, X-ray images of the left hand were centrally assessed by an independent specialist using the Tanner-Whitehouse 2 (RUS) method standardized for Japanese children.
  Height velocity is the yearly height gain. Height velocity SDS for bone age is calculated as following formula; Height velocity SDS = (height velocity - mean) / standard deviation,
  where mean and standard deviation were based on standard Japanese values corresponding to bone age and gender.
  The scores were centred around zero. Negative score indicated a participant was smaller for their age/gender.
Time Frame: Month 12 (at the end of previous study) to 156
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Dose-Increasing Group | Dose-Remaining Group
Number analyzed (Participants) | 29 | 32
SDS
  Month 12 to 24 (Increasing: n=26, Remaining: n=31) | 2.586 (2.268) | 2.461 (1.990)
  Month 24 to 36 (Increasing: n=24, Remaining: n=27) | 1.503 (1.830) | 1.091 (1.852)
  Month 36 to 48 (Increasing: n=22, Remaining: n=22) | 1.196 (1.409) | 0.510 (1.809)
  Month 48 to 60 (Increasing: n=20, Remaining: n=19) | -0.062 (1.775) | 0.913 (2.146)
  Month 60 to 72 (Increasing: n=16, Remaining: n=14) | 0.281 (2.814) | 0.949 (2.729)
  Month 72 to 84 (Increasing: n=13, Remaining: n=13) | -1.249 (2.558) | 0.932 (2.545)
  Month 84 to 96 (Increasing: n=10, Remaining: n=13) | 0.804 (3.440) | 0.286 (2.351)
  Month 96 to 108 (Increasing: n=8, Remaining: n=7) | -0.634 (2.419) | -0.223 (1.352)
  Month 108 to 120 (Increasing: n=5, Remaining: n=5) | 0.070 (4.120) | 0.532 (1.809)
  Month 120 to 132 (Increasing: n=4, Remaining: n=4) | 1.553 (3.019) | 2.718 (0.864)
  Month 132 to 144 (Increasing: n=3, Remaining: n=2) | 2.310 (1.711) | 2.185 (0.304)
  Month 144 to 156 (Increasing: n=2, Remaining: n=0) | 2.710 (2.942) | NA (NA) — Zero participants analyzed at this time point.

6. Secondary Outcome: Height SDS for Bone Age
Description: To measure bone age, X-ray images of the left hand were centrally assessed by an independent specialist using the Tanner-Whitehouse 2 (RUS) method standardized for Japanese children.
  Height SDS for bone age is calculated as following formula; Height SDS = (height - mean) / standard deviation,
  where mean and standard deviation were based on standard Japanese values corresponding to bone age and gender.
  The scores were centred around zero. Negative score indicated a participant was smaller for their age/gender.
Time Frame: Month 12 (at the end of previous study) to 156
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Dose-Increasing Group | Dose-Remaining Group
Number analyzed (Participants) | 29 | 32
SDS
  Month 12 (Increasing: n=27, Remaining: n=31) | -1.19 (1.20) | -0.68 (1.54)
  Month 24 (Increasing: n=26, Remaining: n=31) | -1.15 (1.15) | -0.88 (1.79)
  Month 36 (Increasing: n=24, Remaining: n=27) | -1.20 (1.35) | -1.17 (1.62)
  Month 48 (Increasing: n=22, Remaining: n=22) | -0.74 (1.32) | -1.46 (1.01)
  Month 60 (Increasing: n=20, Remaining: n=19) | -1.16 (1.21) | -1.80 (0.97)
  Month 72 (Increasing: n=16, Remaining: n=14) | -1.78 (1.02) | -1.70 (0.77)
  Month 84 (Increasing: n=13, Remaining: n=13) | -1.85 (1.17) | -2.15 (0.92)
  Month 96 (Increasing: n=10, Remaining: n=13) | -1.77 (1.12) | -2.27 (1.06)
  Month 108 (Increasing: n=8, Remaining: n=7) | -1.41 (0.97) | -1.94 (1.37)
  Month 120 (Increasing: n=5, Remaining: n=5) | -1.58 (1.50) | -1.38 (0.98)
  Month 132 (Increasing: n=4, Remaining: n=4) | -2.10 (1.21) | -0.98 (0.74)
  Month 144 (Increasing: n=3, Remaining: n=2) | -1.40 (0.17) | -0.65 (0.64)
  Month 156 (Increasing: n=2, Remaining: n=0) | -1.55 (0.92) | NA (NA) — Zero participants analyzed at this time point.

ADVERSE EVENTS:
Groups:
- Dose-Remainig Group: Participants in the 0.067 mg/kg/day group in previous study were maintained on the dose in this expention study
Arm/Group | Dose-Increasing Group | Dose-Remainig Group
Serious Adverse Events (participants affected / at risk) | 10/29 | 5/32
Other Adverse Events (participants affected / at risk) | 27/29 | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-Increasing Group (N=29) | Dose-Remainig Group (N=32)
RETINAL DETACHMENT (Eye disorders) | 0 | 1
DEAFNESS (Ear and labyrinth disorders) | 1 | 0
GASTROENTERITIS (Gastrointestinal disorders) | 2 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 | 0
ADENOID HYPERTROPHY (Endocrine disorders) | 1 | 2
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
UPPER RESP TRACT INFECTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HERNIA INGUINAL (Reproductive system and breast disorders) | 1 | 1
OVARIAN DISORDER (Reproductive system and breast disorders) | 1 | 0
HYPOSPADIAS (Congenital, familial and genetic disorders) | 1 | 0
CRYPTORCHISM (Congenital, familial and genetic disorders) | 1 | 0
INFECTION VIRAL (Infections and infestations) | 0 | 1
OTITIS MEDIA (Infections and infestations) | 1 | 1
HEALING IMPAIRED (Infections and infestations) | 0 | 1
INFLICTED INJURY (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-Increasing Group (N=29) | Dose-Remainig Group (N=32)
ACNE (Skin and subcutaneous tissue disorders) | 2 | 3
DERMATITIS (Skin and subcutaneous tissue disorders) | 3 | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 6 | 5
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 2
RASH (Skin and subcutaneous tissue disorders) | 3 | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 2 | 1
RASH PUSTULAR (Skin and subcutaneous tissue disorders) | 4 | 2
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 3 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 2 | 2
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 2
OTITIS EXTERNA (Skin and subcutaneous tissue disorders) | 3 | 2
BULLOUS ERUPTION (Skin and subcutaneous tissue disorders) | 2 | 2
VERRUCA (Skin and subcutaneous tissue disorders) | 1 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 5
HEADACHE (Nervous system disorders) | 4 | 3
CONJUNCTIVITIS (Eye disorders) | 8 | 12
EYE ABNORMALITY (Eye disorders) | 4 | 5
MYOPIA (Eye disorders) | 2 | 0
CONSTIPATION (Gastrointestinal disorders) | 3 | 4
DIARRHOEA (Gastrointestinal disorders) | 5 | 2
VOMITING (Gastrointestinal disorders) | 5 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2
GASTROENTERITIS (Gastrointestinal disorders) | 17 | 10
NAUSEA (Gastrointestinal disorders) | 1 | 2
STOMATITIS (Gastrointestinal disorders) | 2 | 1
TOOTH CARIES (Gastrointestinal disorders) | 4 | 2
TOOTH DISORDER (Gastrointestinal disorders) | 1 | 3
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 2
SGOT INCREASED (Hepatobiliary disorders) | 3 | 1
SGPT INCREASED (Hepatobiliary disorders) | 3 | 1
GLUCOSE TOLERANCE ABNORMAL (Metabolism and nutrition disorders) | 1 | 3
SIALOADENITIS (Endocrine disorders) | 3 | 2
HYPOTENSION POSTURAL (Cardiac disorders) | 2 | 1
COUGHING (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 7 | 9
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 2
RHINITIS (Respiratory, thoracic and mediastinal disorders) | 8 | 12
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 5 | 4
UPPER RESP TRACT INFECTION (Respiratory, thoracic and mediastinal disorders) | 25 | 28
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 9 | 10
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 6 | 6
EOSINOPHILIA (Blood and lymphatic system disorders) | 2 | 3
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 | 4
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 3
LYMPHOCYTES ATYPICA (Blood and lymphatic system disorders) | 2 | 0
PURPURA (General disorders) | 6 | 5
HAEMATOMA (General disorders) | 2 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 2 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 3
OVARIAN DISORDER (Reproductive system and breast disorders) | 3 | 0
SKELETAL MALFORMATION (Congenital, familial and genetic disorders) | 0 | 2
TOOTH MALFORMATION (Congenital, familial and genetic disorders) | 2 | 1
ALLERGIC REACTION (General disorders) | 0 | 3
FEVER (General disorders) | 11 | 1
PAIN (General disorders) | 0 | 2
INFLUENZA-LIKE SYMPTOMS (General disorders) | 16 | 15
INJECTION SITE BLEEDING (Injury, poisoning and procedural complications) | 2 | 0
INFECTION BACTERIAL (Infections and infestations) | 4 | 6
INFECTION VIRAL (Infections and infestations) | 2 | 0
OTITIS MEDIA (Infections and infestations) | 13 | 14
HERPES ZOSTER (Infections and infestations) | 2 | 1
ABSCESS (Infections and infestations) | 0 | 2
VARICELLA (General disorders) | 3 | 2
INFLICTED INJURY (General disorders) | 2 | 4
MOLLUSCUM CONTAGIOSUM (General disorders) | 0 | 2
SCOLIOSIS (General disorders) | 1 | 2
LACERATION (General disorders) | 1 | 3
STING (Injury, poisoning and procedural complications) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.